CLINICAL TRIAL: NCT01578447
Title: Acceptability of Depo-subQ Provera 104 in Uniject Versus Intramuscular Depo-Provera Among HIV-positive Women and Family Planning Providers in Rakai, Uganda
Brief Title: Acceptability of Depo-subQ Provera 104 in Uniject vs. Intramuscular Depo-Provera Among HIV+ Women & Providers, Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Society of Family Planning (Other); Bill and Melinda Gates Foundation (Other); Rakai Health Sciences Program (Other)
Responsible Party: Principal Investigator, Ronald Gray, Professor, Johns Hopkins Bloomberg School of Public Health
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 00003213
Record Dates: First submitted 2012-04-04; First posted 2012-04-17 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Acceptability of Different Contraceptive Injection Types
Keywords: injectable contraception; acceptability; intramuscular; subcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Depo-SubQ Provera 104 in Uniject (Other)
  Interventions: Drug: DepoSubQ Provera 104 in Uniject
- Intramuscular DMPA (Other)
  Interventions: Drug: Intramuscular DMPA

INTERVENTIONS:
Drug: DepoSubQ Provera 104 in Uniject — DepoSubQ Provera 104 in Uniject
  Arms: Depo-SubQ Provera 104 in Uniject
Drug: Intramuscular DMPA — Intramuscular DMPA
  Arms: Intramuscular DMPA

SUMMARY:
The purpose of this study is to assess acceptability and side effects of a low-dose injectable contraceptive formulation which is delivered under the skin (subcutaneously), as compared with injectable contraception delivered into the muscle (intramuscularly) among adult HIV-positive women who attend mobile clinics for HIV care and wish to use injectable contraception. The investigators will also assess experiences experiences delivering these two types of injections among health care providers working within the HIV care clinics.

ELIGIBILITY:
Inclusion Criteria:

* HIV+
* Woman aged 18-45
* Wishes to prevent pregnancy by use of injectable contraception and intends to continue using injectable contraception for next nine months
* Medically eligible for injectable contraception
* Capable of providing informed consent
* Willing to provide contact information
* Agrees to trial participation
* Intends to live in the area for the next nine months
* May or may not be currently using a first-line antiretroviral therapy regimen (includes: AZT/3TC/EFV; AZT/3TC/NVP; CBV/EFV; D4T/3TC/EFV; D4T/3TC/NVP; TDF/3TC/EFV; TDF/3TC/NVP)

Exclusion Criteria:

* Currently pregnant
* Desires pregnancy within next nine months
* Contraindications to using injectable contraception
* On second-line antiretroviral therapy regimen

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 356 (Actual)
Dates: Start 2012-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Preferred injection method | 6 months
  Preference for subcutaneous injection, intramuscular injection, or no preference between the two

SECONDARY OUTCOMES:
Acceptability, satisfaction, and problems encountered with subcutaneous injection versus intramuscular injection, as reported by HIV/family planning care providers | Baseline, 10 months
  E.g., problems encountered, preference to give more, same amount, or fewer of each kind of injection, advantages and disadvantages of each kind of injection, difficulty of administration, perception of client experience, which type of injectable prefers to administer, whether preferences are impacted by HIV status of client
Hypothetical acceptability of contraceptive injections provided by community health care worker, trained and trusted friend or family member, or self-administration | Baseline, 3 months, 6 months
  In this study, all injections will be provided by a trained medical professional, but we will ask women if they would hypothetically find provision by community health workers, a trained trusted friend or family member, or self-administration acceptable
Pregnancy incidence | 3 months, 6 months
  Will not be compared according to study product, since all participants will utilize both products in this crossover trial.
Side effects | Baseline, 3 months, 6 months
  Including pain/injection/soreness at injection site and other reported side effects
Continuation of use of injectables | 3 months, 6 months
  Proportion of enrolled women who continue using injectable contraception at follow up visits
Future use intentions | Baseline, 3 months, 6 months
  Whether plans to use injectable contraception again in three months
Likelihood of recommending method to a friend | Baseline, 3 months, 6 months
  How likely participant would be to recommend this contraceptive method to a friend
Level of satisfaction with method | Baseline, 3 months, 6 months
  Level of satisfaction with method of contraception injection received

CONTACTS AND LOCATIONS:
Overall Officials: Ron H Gray, MD, MSC, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Rakai Health Sciences Program, Kalisizo, Uganda

REFERENCES:
- [Result] Polis CB, Nakigozi GF, Nakawooya H, Mondo G, Makumbi F, Gray RH; Members of the Rakai Health Sciences Program Sayana Press study team. Preference for Sayana(R) Press versus intramuscular Depo-Provera among HIV-positive women in Rakai, Uganda: a randomized crossover trial. Contraception. 2014 May;89(5):385-95. doi: 10.1016/j.contraception.2013.11.008. Epub 2013 Nov 15. PMID 24332432